CLINICAL TRIAL: NCT02105168
Title: Identification of Marker of Primary or Acquired Resistance to Anti Tumorous Treatment in Patients With Lung Cancer or Melanoma
Brief Title: Identification of Marker of Primary or Acquired Resistance to Anti Tumorous Treatment
Acronym: MSN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2008-A00373-52; 2007/1363 (Other: CSET number)
Record Dates: First submitted 2014-03-31; First posted 2014-04-07 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Melanoma; Non Small Cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental arm (Experimental): Blood sample Tumorous biopsy Healthy material sample
  Interventions: Procedure: Blood sample; Procedure: Tumorous biopsy; Procedure: Healthy material sample

INTERVENTIONS:
Procedure: Blood sample — Optional
Procedure: Tumorous biopsy — Optional
Procedure: Healthy material sample — Optional

SUMMARY:
Lung Cancer and melanoma relapsed frequently whereas its very sensitive to treatment such as chemotherapy or radiotherapy. The purpose of this study is to have a better understanding of why those patients are relapsing using next generation sequencing to identify rare mutations and assessed their predictive value.

ELIGIBILITY:
Inclusion Criteria:

1. Cytological or histological diagnosis of SCLC, NSCLC or melanoma
2. Patients age >/= 18 years old
3. Indication of treatment using platinum salts for lung cancer except for patient with NSCLC treated by surgery for whom platinum salts is not indicated
4. If a biopsy is proposed, lesion lust be easily accessible
5. Signed informed consent

Exclusion Criteria:

1. Patients unable to follow the protocol
2. Consent refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2009-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Mutation rate on tumorous material | Assessed at the time of inclusion
  Assessed at the time of inclusion using tumorous material used for diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Besse, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val de Marne, France

REFERENCES:
- [Derived] Mezquita L, Preeshagul I, Auclin E, Saravia D, Hendriks L, Rizvi H, Park W, Nadal E, Martin-Romano P, Ruffinelli JC, Ponce S, Audigier-Valette C, Carnio S, Blanc-Durand F, Bironzo P, Tabbo F, Reale ML, Novello S, Hellmann MD, Sawan P, Girshman J, Plodkowski AJ, Zalcman G, Majem M, Charrier M, Naigeon M, Rossoni C, Mariniello A, Paz-Ares L, Dingemans AM, Planchard D, Cozic N, Cassard L, Lopes G, Chaput N, Arbour K, Besse B. Predicting immunotherapy outcomes under therapy in patients with advanced NSCLC using dNLR and its early dynamics. Eur J Cancer. 2021 Jul;151:211-220. doi: 10.1016/j.ejca.2021.03.011. Epub 2021 May 19. PMID 34022698